CLINICAL TRIAL: NCT03569124
Title: Interpretation of Endoscopic Characteristics of Colorectal Polyps With Blue Light Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Midwest Biomedical Research Foundation (Other)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Chair, Department of Gastroenterology, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: 00983
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Identification of Colorectal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training group
  Interventions: Other: Teaching tool for identification of colorectal polyps
- Non-Training group

INTERVENTIONS:
Other: Teaching tool for identification of colorectal polyps — This is a teaching session on how to identify the colorectal polyps shot in blue light imaging.
  Groups: Training group

SUMMARY:
Interpretation of endoscopic characteristics of colorectal polyps with Blue Light Imaging A study of BLI images and videos of colorectal polyps will be presented initially as a training set followed by with explanation and teaching in a didactic session to two separate groups. A post-test will be conducted to look at the quality of the learning experience.

To evaluate the teaching tool regarding the criteria for BLI images of colorectal polyps by the following measures

* Inter-observer agreement between same and different groups
* Accuracy in describing the morphology of colorectal polyps • This new teaching tool will improve
* Inter-observer agreement by at least 5%- 10% (depending on the group)
* Accuracy by at least 5%- 10% (depending on the group)• To determine the improvement of inter-observer agreement in identifying/ describing colorectal polyps after the didactic session in both the groups
* Overall Accuracy, Sensitivity, Specificity, Positive predictive value and negative predictive value pre-and post-test in both the groups

ELIGIBILITY:
Inclusion Criteria All gastroenterology attending physicians, gastroenterology fellows, residents and medical students at the VA medical center

Exclusion Criteria Not willing to participate H/O colour blindness or visual impairment Any intellectual disability

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants are contacted while they are at the VA medical centre. All gastroenterology attending physicians, gastroenterology fellows, residents and medical students will be notified about the study and asked about the willingness to participate if they fit the inclusion/exclusion criteria. Practicing gastroenterologists and trainees will be contacted and inquired about their intent of participating in the assessment of images/videos. This is a voluntary project and not a part of any mandatory training. There is no coercion of participants who do not want to participate.
  This study includes only the images and videos from standard pre-existing database. This database was developed by European investigators for educational purposes. This information has no patient identifiable parameters. This information is stored in a secure server with guarded access.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
inter-observer agreement in identifying/ describing colorectal polyps | 1 year
  it is measured by kappa statistic which measures the agreements of the total interpretations

SECONDARY OUTCOMES:
Accuracy | 1 year
  Accuracy comparison between training and non training groups
Sensitivity | 1 year
  Sensitivity comparison between training and non training groups
Specificity | 1 year
  Specificity comparison between training and non training groups
Positive predictive value | 1 year
  Positive predictive value comparison between training and non training groups
Negative predictive value | 1 year
  Negative predictive value comparison between training and non training groups

IPD SHARING:
Plan to Share IPD: No
No need of sharing as the participants are the institutional ones

REFERENCES:
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Background] Rastogi A, Keighley J, Singh V, Callahan P, Bansal A, Wani S, Sharma P. High accuracy of narrow band imaging without magnification for the real-time characterization of polyp histology and its comparison with high-definition white light colonoscopy: a prospective study. Am J Gastroenterol. 2009 Oct;104(10):2422-30. doi: 10.1038/ajg.2009.403. Epub 2009 Jul 7. PMID 19584829
- [Background] Togashi K, Nemoto D, Utano K, Isohata N, Kumamoto K, Endo S, Lefor AK. Blue laser imaging endoscopy system for the early detection and characterization of colorectal lesions: a guide for the endoscopist. Therap Adv Gastroenterol. 2016 Jan;9(1):50-6. doi: 10.1177/1756283X15603614. PMID 26770267